CLINICAL TRIAL: NCT03519165
Title: Restrictive or Individualized Goal-Directed Fluid Replacement Strategy in Ovarian Cancer Cytoreductive Surgery- A Prospective Randomized Controlled Trial
Brief Title: Restrictive or Individualized Goal-Directed Fluid Replacement Strategy in Ovarian Cancer Cytoreductive Surgery
Acronym: RIGoROCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC/TMC/56/15
Record Dates: First submitted 2016-03-22; First posted 2018-05-08 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; goal-directed fluid therapy; SVV
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Flotrac System 4.0 Edwards Lifesciences, Irvine, CA, USA
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Group C) (No Intervention): Conventional Fluid therapy guided by clinical parameter
  Intraoperative fluid therapy will include maintenance fluid and replacement of the surgical loss. Aim to maintain MAP > 65 mmHg, CVP 8-12 cm H2O and urine output > 0.5 ml/kg/h.
- Goal directed group (Group G) (Active Comparator): Intervention: Machine guided fluid therapy using EV1000 (FloTrac System 4.0 Edward Lifesciences, Irvine, CA, USA)
  Intraoperative fluid therapy will be targeted to SVV <13%, SVI > 35ml/m2/ beat, SVRI more than equal to 1900 dynes-sec/cm-5/m2 using EV1000 floTrac monitor in addition to clinical parameters like MAP, CVP and urine output
  Interventions: Device: EV1000(FloTrac System 4.0)

INTERVENTIONS:
Device: EV1000(FloTrac System 4.0)
  Arms: Goal directed group (Group G)

SUMMARY:
This is a single center prospective randomized controlled study comparing the postoperative outcome after cytoreductive surgery in ovarian cancer patient after using restrictive or individualized goal-directed fluid replacement strategy (GDT). Aim of this study will be to test the hypothesis that intra-operative SVV-guided fluid optimization during ovarian cancer cytoreductive surgery:

1. reduces the postoperative length of hospital stay,
2. cost-effective,
3. GDT will be more beneficial in cases of PDS compared to IDS or cytoreductive procedures of shorter duration.
4. GDT improves intraoperative tissue perfusion/ oxygenation and improves immediate postoperative morbidity.

Intra-operatively fluid of choice in both groups will be lactate-free crystalloid at 1.0 ml/kg/h for maintenance and gelofusine for fluid bolus of 3ml/kg over 5 minutes. In group C intraoperative fluid therapy will include maintenance fluid and replacement of the surgical loss. Aim will be to maintain MAP > 65 mmHg, CVP 8-12 cm H2O and urine output > 0.5 ml/kg/h. In group G intraoperative fluid therapy will be targeted to SVV <13%, SVI > 35ml/m2/ beat, SVRI more than equal to 1900 dynes-sec/cm-5/m2 in addition to clinical parameters like MAP, CVP and urine output.

Primary outcome will be length of hospital stay (LOS). Secondary outcomes will be cost of surgical treatment episode (admission till fit to discharge), postoperative morbidity survey (POMS) and 30 day morbidity and mortality.

DETAILED DESCRIPTION:
Aims & objectives:

The purpose of the study is to test the hypothesis that intra-operative SVV-guided fluid optimization during ovarian cancer cytoreductive surgery -

1. Reduces the postoperative length of hospital stay.
2. GDT is more cost-effective.
3. GDT will be more beneficial in cases of PDS compared to IDS.
4. GDT reduces postoperative morbidity.

Justification for study:

Cytoreductive surgery in ovarian cancer is usually associated with significant fluid shift attributable to suboptimal nutritional status, prolonged preoperative starvation, intraoperative blood and fluid loss, pharmacological vasodilation by neuraxial (epidural) and systemic anaesthetic drugs, intraoperative evaporative loss and the vasodilation due to systemic inflammatory response to surgery (SIRS), which was comparatively more in case of ovarian surgery. This results in hypotension and altered hemodynamics in the intra-operative and immediate

post-operative settings and the need for rigorous hemodynamic monitoring in the perioperative period. Among 3 different strategies, liberal or conservative one is associated with risk of overhydration, whereas restrictive therapy can cause hypoperfusion and related complications. A goal-directed fluid therapy has been shown to optimise intravascular volume in major abdominal surgery, which is the key determinant of cardiac output and oxygen delivery to tissues. This strategy results in use of more advanced hemodynamic monitors and increased costs thereof, and possibly, more total fluid requirements. A restrictive fluid strategy targeting physiological parameters alone, utilizes less costly modalities of monitoring and less overall fluid infused. But total healthcare cost associated with reduced rate of complications and thereby less hospital stay can neutralize that extra-cost of advanced monitoring (approximately Rs 8,000 per patient for consumables) and become more cost effective. The current standard of care in Tata Medical Center (TMC) has been a fluid therapy guided by clinical parameters. Although there is strong evidence supporting goal-directed approach to perioperative fluid therapy in case of major abdominal surgery, which has also been incorporated in enhanced recovery protocol and adopted worldwide, there is no such evidence for gynaec-oncological surgery, especially in ovarian cancer. So, investigators would like to conduct the proposed study to find-out the optimal fluid management strategy for ovarian cytoreductive surgery. As previously mentioned, investigators' data might indicate that the standard approach may lead to tissue hypoperfusion and approximately 2-3 liters of deficit which needs replacement under monitoring in order to avoid fluid overload.

Arguably, all patients of major cytoreductive surgery should require goal directed therapy and therefore randomization can potentially harm a subset of patients who would then receive restricted therapy instead of goal directed therapy. However, the standard regimen which is currently used in our setting is restrictive and SVV is also being increasingly used routinely only at the clinician's discretion including in ovarian cancer cases. Therefore no harm is anticipated from this intervention in either group. The only implication is of cost and resources; goal directed therapy has resource implications- both in terms of availability of machine and additional cost to the patient due to the consumables. A non-randomized prospective observational study would be feasible but will not be able to select which patients would benefit maximum from GDT due to selection bias. Therefore, a randomized study may help to identify a select group of patients who might benefit the maximum and therefore SVV directed fluid administration could be further stratified to be cost-effective due to reduction of postoperative length of hospital stay and morbidity.

From personal communication investigators know that, 3 trials of perioperative fluid therapy are ongoing now in India. Out of those 3 trials, 2 are in abdominal surgery and one is in hyperthermic intraperitoneal chemotherapy (HIPEC) surgery. Other cancer centers expressed interest to undertake similar trial in ovarian cytoreductive surgery. Therefore investigators may collaborate with other centers in future for a larger study based on the results; however, at present a single institutional study will be conducted to minimize bias associated with heterogeneity in surgical practice on cytoreduction.

Benefit:

This study will help investigators to guide fluid therapy in the perioperative period in ovarian cancer patients undergoing cytoreductive surgeries. This study should also help to find a strategy to prevent both fluid overload as well as under filling to avoid hypo perfusion and organ damage in this vulnerable group of patients. This strategy can even be adopted in other patient populations undergoing colorectal, hepatobiliary, thoraco-abdominal and HIPEC surgeries. These data will also inform whether a stratified approach can be adopted to selectively use SVV monitoring according to the predicted surgical complexity, type of cytoreduction and duration of surgery to optimize resources and improve cost-effectiveness.

Risks This study will utilize an existing technology, which is already in use. Therefore SOPs will be followed including reporting of adverse events, monitoring, documentation and safety reporting. The intervention is fluid bolus guided by advanced haemodynamic parameters (EV1000 monitor). Therefore risks are theoretical only. Risks related to the invasive procedures are same in both arms, which include pneumothorax, haemothorax, haemo-pneumothorax, bleeding, catheter-related infection and peripheral ischemia.

Methodology:

Site of Study OT complex and Intensive Care Unit, Department of Anaesthesiology & Critical Care, Tata Medical Center, Kolkata

Study Structure Design:

Prospective randomized controlled trial - Patients and assessors will be blinded.

Population: All ovarian cancer patients undergoing major debulking surgery at TMC Kolkata (except- completion staging).

Sample size:

The study design was based on a retrospective audit at TMC that found the current median postoperative length of stay to be 10 days after cytoreductive surgery in ovarian cancer. To detect a reduction of 2 post-operative days with median postoperative length of stay to be 10 days in the restrictive group and 8 days in the goal directed group with a SD=3 days for 80% power at a significance level of 0.05, 37 patients are needed in each group (Total=74). As there is a difference in the median postoperative length of stay between the PDS and IDS group as mentioned earlier, at least 20 patients in each of the IDS and PDS groups would be needed for both the goal directed and restrictive group.

So the study would continue till each of the four combinations: Goal Directed (IDS), Goal Directed (PDS), Control (IDS) and Control (PDS) have at least 20 patients. To account for possible 10% attrition rate/ loss to follow up, 44 patients would be required in each group

Method of Randomization:

In addition to having higher median LOS in hospital, patients undergoing PDS are more likely to have ascites, major peritoneal stripping, higher surgical complexities and intraoperative fluid loss. Therefore, pre-randomization stratification will be done for type of surgery. Patients would be enrolled separately into PDS and IDS groups. Then for each group, patients would be randomized to get the standard or the goal directed therapy mentioned in the sealed envelopes based on computer generated random numbers.

After randomization and inclusion into a study arm, patients will be excluded in an event of the following: the procedure is abandoned/ open and close, duration of procedure is less than 4 hours, and any critical incident during operation (i.e. major blood loss/ medical condition/ shock) requiring intense fluid resuscitation. Following factors will be analyzed for univariate and multivariate analysis: ASA status, duration of surgery in minutes, surgical complexity score, intraoperative fluid loss, total vs. partial peritonectomy, comorbidities (Possum-P), massive blood loss and transfusion. Analysis will be on a per protocol basis as well as intention to treat.

Blinding:

* As the envelope would be opened after induction of GA, the patient will be blinded to the group she is allocated to.
* Post operative data will be collected by the ICU Consultant/ medical officer and Gynaec-oncosurgery team, who would not be part of the study and unaware about the allocation will follow up patients and decide on fitness to discharge. Outcome will also be verified according to predefined criteria by other clinicians from Gynaec-oncosurgery team, who are not aware about the allocated study group.

Statistical Analysis:

All statistical analyses and all summary tables and listings will be prepared using SASÒ release 8.3 or higher (SAS Institute, Inc., Cary, NC). Standard descriptive summaries will include the N, mean, median, standard deviation, minimum and maximum for continuous variables, and the number and percent for categorical variables. All statistical test of comparison will be based on 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Cytoreductive surgery for ovarian cancer-

  * PDS: primary (chemo-naïve patients including completion staging/ primary debulking and secondary cytoreduction)
  * IDS: interval debulking surgery (after chemotherapy)
* American Society of Anesthesiology (ASA-PS) score of 1 - 3
* Age more than 18 years and less than 65 years
* Surgery of duration more than 240 minutes
* Presumed blood loss more than 500 ml
* Elective surgery

Exclusion Criteria:

* Patient refusal
* Inability to give consent
* Laparoscopic surgery, Emergency surgery, patients undergoing HIPEC
* Age younger than 18 years & more than 65 yrs, BMI > 40
* Patients with LVEF < 30%, Arrhythmia, Acute MI (within 30 days)
* COPD with FEV1 < 50%
* Coagulopathy (platelet <50000/μL, aPTT > x2 control, INR >1.5)
* Significant liver dysfunction (liver enzymes >x3 times normal)
* Significant renal dysfunction (creatinine >x2 times normal)
* Psychiatric disorders
* Sepsis or SIRS
* Hypersensitivity to Gelofusine

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Postoperative length of Stay (LOS) in hospital in days | through study completion, an average of 2 years
  From day of surgery to the day of fit to discharge

SECONDARY OUTCOMES:
Cost of treatment | through study completion, an average of 2 years
  cost of treatment includes direct medical cost and out of pocket expenditure
Post operative morbidity survey (POMS survey) | on 1,3,5 and 7th postoperative day and through study completion, an average of 2 years
  The postoperative morbidity survey (POMS) is a nine-domain (Pulmonary, infection, renal, GIT, CVS, Neurological, haematological, wound and pain) system that prospectively identifies short-term morbidity after surgery. For each of the nine domains morbidity is recorded on the presence or absence of preset criteria.(PubMed ID: 10439777)
30 day morbidity and mortality | through study completion, an average of 2 years
  No. of patients in each group with grade 3 to 5 postoperative complications (Clavien-Dindo Classification) and description of complication

CONTACTS AND LOCATIONS:
Overall Officials: Jyotsna Goswami, MD, Principal Investigator — Tata Medical Center; Asima Mukhopadhyay, MD, PHD, Principal Investigator — Tata Medical Center
Locations (1):
- Tata Medical Centre, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McKenny M, Conroy P, Wong A, Farren M, Gleeson N, Walsh C, O'Malley C, Dowd N. A randomised prospective trial of intra-operative oesophageal Doppler-guided fluid administration in major gynaecological surgery. Anaesthesia. 2013 Dec;68(12):1224-31. doi: 10.1111/anae.12355. Epub 2013 Sep 30. PMID 24116747
- [Background] Chattopadhyay S, Mittal S, Christian S, Terblanche AL, Patel A, Biliatis I, Kucukmetin A, Naik R, Galaal K. The role of intraoperative fluid optimization using the esophageal Doppler in advanced gynecological cancer: early postoperative recovery and fitness for discharge. Int J Gynecol Cancer. 2013 Jan;23(1):199-207. doi: 10.1097/IGC.0b013e3182752372. PMID 23154265
- [Background] Bennett-Guerrero E, Welsby I, Dunn TJ, Young LR, Wahl TA, Diers TL, Phillips-Bute BG, Newman MF, Mythen MG. The use of a postoperative morbidity survey to evaluate patients with prolonged hospitalization after routine, moderate-risk, elective surgery. Anesth Analg. 1999 Aug;89(2):514-9. doi: 10.1097/00000539-199908000-00050. PMID 10439777